CLINICAL TRIAL: NCT05532735
Title: Open-label, Dose Ascending Safety, Tolerability, and Proof of Concept Study to Evaluate the Use of ANXV (Human Recombinant Annexin A5) in the Treatment of Subjects With Recently Diagnosed Retinal Vein Occlusion
Brief Title: Safety and Proof of Concept Study of ANXV (Annexin A5) in Patients With Retinal Vein Occlusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annexin Pharmaceuticals AB (Industry)
Collaborators: InFocus Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANN-004
Record Dates: First submitted 2022-07-18; First posted 2022-09-08 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 2 mg ANXV (Experimental): ANXV (human recombinant Annexin A5), infusion, 2 mg daily during five days.
  Interventions: Biological: ANXV
- 4 mg ANXV (Experimental): ANXV (human recombinant Annexin A5), infusion, 4 mg daily during five days.
  Interventions: Biological: ANXV
- 1 mg ANXV (Experimental): ANXV (human recombinant Annexin A5), infusion, 1 mg daily during five days.
  Interventions: Biological: ANXV
- 6 mg ANXV (Experimental): ANXV (human recombinant Annexin A5), infusion, 6 mg daily during five days.
  Interventions: Biological: ANXV
- 8 mg ANXV (Experimental): ANXV (human recombinant Annexin A5), infusion, 8 mg daily during five days.
  Interventions: Biological: ANXV

INTERVENTIONS:
Biological: ANXV — ANXV (Human recombinant Annexin A5 protein)

SUMMARY:
Open-label, dose ascending safety, tolerability, and proof of concept study to evaluate the use of ANXV (human recombinant Annexin A5) in the treatment of subjects with recently diagnosed Retinal Vein Occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated), and any authorizations required by local law and be able to comply with all study requirements
2. Male or female, ≥18 years of age at the time of informed consent
3. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., ≥6 weeks post bilateral salpingectomy, bilateral oophorectomy with or without hysterectomy) or post-menopausal (12 months of spontaneous amenorrhea in females > 55years of age or, in females ≤55 years, or 12 months of spontaneous amenorrhea without an alternative medical, or 12 months with an elevated Follicle Stimulating Hormone (FSH) level Males must either be surgically sterile or abstinent*, or if engaged in sexual relations with a female of child-bearing potential, the subject or the subject's non-pregnant female partner must use a highly effective contraception method from the time of signing the Informed Consent Form (ICF) until at least 30 days after the last dose of study drug; Refer to Section 10.3 for acceptable methods

   *Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods). Declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception (Section 10.3).
4. Onset of symptoms of Retinal Vein Occlusion within 23 days prior to informed consent
5. The criterion has been removed
6. The criterion has been removed
7. Clear ocular media and adequate pupillary dilation in the Study Eye to permit high quality retinal imaging
8. Willing to refrain from strenuous exercise/activity (for example heavy lifting, weight training, intense aerobics classes etc.) for at least 72 hours prior to study visits
9. A negative rapid SARS-CoV-2 (COVID) test on Day 1 prior to initiation of study drug infusion

Exclusion Criteria:

Subjects will not be eligible if they have any of the following criteria:

Study Eye only:

1. A severe (≥0.9 log, Grade 3+ or worse) Relative Afferent Pupillary Defect (RAPD)
2. Evidence of deep intraretinal hemorrhage involving the center 1mm of the macula
3. Evidence of neovascularization
4. Ocular disorders/additional eye disease, which in the opinion of the Investigator may confound interpretation of study results, compromise protocol assessments or are likely to require intervention during the study, including, but not limited to, atrophy of the retinal pigment epithelium, sub-retinal fibrosis, organized hard exudate plaque, clinically significant diabetic macular edema, retinal detachment, macular hole, vitreomacular traction, macular epiretinal membrane, clinically significant cataract, vitreal opacities or hemorrhage, glaucoma with documented visual field loss, ischemic optic neuropathy, retinitis pigmentosa or choroidal neovascularization of any cause (e.g., Age-related Macular Degeneration (AMD), ocular histoplasmosis, toxoplasmosis, or pathologic myopia)
5. Laser photocoagulation in the study eye within the preceding 6 months prior to the Screening Visit
6. Receipt within the past 6 months prior to the Screening Visit of any intraocular surgery (including refractive surgery, cataract surgery), or intravitreal (IVT) injection, or planned intraocular surgery or procedure during the study, unless approved by Medical Monitor or Sponsor
7. Recent (6 months) history, or current evidence of ocular herpetic diseases (including herpes simplex virus, varicella zoster or cytomegalovirus), unless approved by Medical Monitor or Sponsor

   Fellow Eye:
8. BCVA in the Fellow eye of ≤70 ETDRS letters (approximately 20/40 or less), unless approved by the Medical Monitor or the Sponsor

   Both Eyes:
9. Within 6 months prior to the Screening Visit, use of medications known to be toxic to the retina, lens, or optic nerve (e.g., desferoxamine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, and ethambutol)
10. Known hypersensitivity or allergy to fluorescein (e.g., bronchospasm, rash, etc.) or to any component of the study products or a contraindication to dilation of the pupil or fixed pupils; mild allergies without angio-edema or treatment need may be acceptable if deemed not to be of clinical significance (including but not limited to allergy to animals or mild seasonal hay fever)
11. An IOP greater than 24 mmHg that is not controlled with medication or surgery at the time of the Screening Visit
12. Recent (6 months) history of, or presence of uveitis, presence of intraocular inflammation (history of blepharitis is not exclusionary), current ocular infection

    General:
13. Unwillingness or inability to attend all study visits and/or perform all procedures/tests/examinations, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator
14. Any medical or surgical procedure or trauma within 4 weeks prior to the day of Treatment 1 (study drug administration), or planned major surgery within the duration of the study through Day 120, unless approved by Medical Monitor or Sponsor
15. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
16. Prior exposure to a recombinant Annexin A5
17. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to biologics (for example systemically administered recombinant proteins/peptides; a similar drug class to ANXV)
18. Uncontrolled hypertension (systolic > 180 mmHg or diastolic > 110 mmHg)
19. Current use of any systemically administered anti-angiogenic agent (e.g., bevacizumab, sunitinib, cetuximab, sorafenib, pazopanib) or corticosteroids, approved or 5 half-lives of investigational agent
20. Diagnosed untreated systemic metastasis malignancy
21. A current systemic infection or inflammation that may require antiviral or antimicrobial therapy that will not be completed prior to Screening Visit, or that in the opinion of the Investigator and with concurrence of the Medical Monitor may either put the subject at risk or may influence the results of the study, or the subject's ability to participate in the study
22. Treatment with another investigational drug, biological agent, or device within 3 months of Screening Visit, or 5 half-lives of investigational agent, whichever is longer or planned participation in an investigational trial from signing ICF through Day 120
23. History of thromboembolic events or deep venous thrombosis within 3 months of Screening Visit
24. Current use of anticoagulant medication (any medications that might have effect on coagulation, hemostasis, and platelets); low dose aspirin allowed prior to informed consent but must be stopped at the time of consent; may begin again 1 day post Treatment 5 infusion
25. Current daily use of benzodiazepines (intermittent use permissible with Medical Monitor or Sponsor approval)
26. Clinically significant abnormal coagulation parameters at baseline
27. The criterion has been removed from the protocol
28. History of autoimmune disease with anticipated presence of persistent Annexin A5 antibodies, e.g., antiphospholipid syndrome, systemic lupus erythematosus, rheumatoid arthritis, Behcet disease or systemic sclerosis
29. Inherited blood disorder (e.g. sickle cell disease, thalassemia)
30. History of unstable coronary artery disease or cerebrovascular accident within the last 3 months
31. GFR below 70 mL/min at baseline
32. Current drug or alcohol abuse, current excessive smoking (i.e., ≥ 20/day)
33. Known history of or positive test for hepatitis C or chronic hepatitis B
34. Class III obesity (Body Mass Index ≥ 40kg/m2), at the time of informed consent (Sponsor may accept eligibility for a subject with higher Body Mass Index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Safety - Treatment Emergent Adverse Events | 120 days
  Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Safety - Anti-drug antibodies | 120 days
  Incidence and titer of anti-drug antibodies (ADA) to ANXV pre- and post-administration

SECONDARY OUTCOMES:
Safety - Slit lamp | 120 days
  Slit-lamp biomicroscopy including intraocular pressure (IOP) and dilated indirect ophthalmoscopy
Safety - Gonioscopy | 120 days
Safety - Best Corrected Visual Acuity (BCVA) | 120 days
  Distance BCVA by manifest refraction should be performed utilizing the ETDRS chart at a starting distance of 4 meters
Safety - laboratory parameters | 15 days
  Concentration of analytes in Chemistry panel, lipid panel, hematology, coagulation, inflammatory and urinalysis
Safety - vital signs Blood Pressure | 15 days
  Blood pressure (BP)
Safety - vital signs Heart rate | 15 days
  Heart rate (HR)
Safety - vital signs Weight | 15 days
  Weight
Safety - vital signs Body Temperature | 15 days
  Body temperature
Safety - vital signs Respiratory rate | 15 days
  Respiratory rate (RR)
Safety - vital signs Pulse oximetry | 15 days
  Pulse oximetry
Safety - ECG | 15 days
  12-lead ECG
Safety - ANXV anti-drug antibodies Persistence | 12 months
  Persistence anti-drug antibodies
Safety - ANXV anti-drug antibodies Titer | 12 months
  Titer of anti-drug antibodies
Efficacy - Microperimetry Change from baseline | 120 days
  Change from baseline in microperimetry mean retinal sensitivity calculated on all stimulus points ≤20 dB at baseline (MSEff), at Days 8, 15, and 29
Efficacy - Microperimetry Stimulus points | 120 days
  Number of microperimetry stimulus points that improve by ≥7decibels (dB) from baseline to Day 8 and 29 after the first ANXV infusion
Efficacy - Microperimetry Improvement over baseline | 120 days
  Number of subjects with an improvement over baseline in MSEff of ≥7dB at Days 8, 15 and 29 (MMP positive responders, MMP-pos)
Efficacy - Microperimetry Incremental loss | 120 days
  Number of subjects with an incremental loss over baseline in MSEff of ≥7dB at Days 8, 15 and 29 (MMP negative responders, MMP-neg)
Efficacy - Microperimetry Improvement of ≥7dB | 120 days
  Number of subjects with an improvement of ≥7dB over baseline in ≥5 stimulus points at Days 8, 15 and 29 (MMP positive-5 responders, MMP-pos-5)
Efficacy - Microperimetry MMP negative-5 responders | 120 days
  Number of MMP negative-5 responders, i.e., subjects with an incremental loss over baseline of ≥7dB in ≥5 stimulus points at Days 8, 15 and 29 (MMP-neg-5)
Efficacy - BCVA Improvement | 120 days
  Number of subjects with an improvement of ≥15 ETDRS letters over baseline at Days 8, 15 and 29
Efficacy - BCVA Improvement or letter score ≥78 | 120 days
  Number of subjects with an improvement of ≥15 ETDRS letters over baseline or an ETDRS letters score ≥78 at Days 8, 15 and 29
Efficacy - Spectral Domain Optical Coherence Tomography / Spectral Domain Optical Coherence Tomography Angiography (SD-OCT/OCTA) SD-OCT | 120 days
  Change from baseline in Center Subfield Macular Thickness (CMT), Macular Volume and Outer Nuclear Layer (ONL) thickness on SD-OCT at Days 8, 15 and 29
Efficacy - Spectral Domain Optical Coherence Tomography / Spectral Domain Optical Coherence Tomography Angiography (SD-OCT/OCTA) OCTA | 120 days
  Change from baseline in Foveal Avascular Zone (FAZ) and Vessel Density (VD) on OCTA at Days 8, 15 and 29
Efficacy - Ultra-Wide Field Fluorescein Angiography (UWF-FA) Size of Retinal Area of Non-Perfusion | 120 days
  Change from baseline at Days 8 and 29 in the size of Retinal Area of Non-Perfusion (RANP) for:
  1. all the retina captured by UWF-FA
  2. in posterior pole
Efficacy - Ultra-Wide Field Fluorescein Angiography (UWF-FA) Conversion from non-ischemic RVO to ischemic RVO | 120 days
  Number of subjects at Days 8, and 29 with:
  1. RANP ≥30 DA
  2. RANP ≥10 DA Rate of conversion from non-ischemic RVO (niRVO) to ischemic RVO (iRVO) by Day 29
Efficacy - Need for rescue treatment with anti Vascular Endothelial Growth Factor (aVEGF) therapy | 29 days
  Number of subjects requiring rescue with an aVEGF by Day 29
Ischemic Index | 120 Days
  Change in Ischemic Index (ISI) from baseline at Days 8 and 29
Pharmacokinetic (PK) profile | 5 days
  ANXV concentration on Days 1 and 5 pre-infusion and at 15, 30, and 40 minutes and 1, 1.5, 2 and 3.5 hours after the start of the infusion

OTHER OUTCOMES:
ANXV binding sites | 43 days
  Assessment of ANXV binding sites (PS on circulating cells and microparticles) in whole blood sample, Day 1 (pre- infusion), Days 1 and 5 at 5 minutes post infusion, and 3 hours post end of infusion and on Days 8, 15 and 43
Endogenous Annexin A5 | 43 days
  Endogenous Annexin A5 levels, Day 1 (pre-infusion) and Days 8, 15 and 43

CONTACTS AND LOCATIONS:
Overall Officials: Anna Frostegård, Study Director — Annexin Pharmaceuticals
Locations (7):
- United States (7):
  - Eye Associates of Northeast Louisiana, West Monroe, Louisiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Retina Consultants of Texas, Bellaire, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Virginia Retina Center, Warrenton, Virginia

IPD SHARING:
Plan to Share IPD: No